CLINICAL TRIAL: NCT04339816
Title: Azithromycin Added to Hydrochloroquine in Patients Admitted to Intensive Care Due to Coronavirus Disease 2019 (COVID-19)- Randomised Controlled Trial
Brief Title: Azithromycin Added to Hydrochloroquine in Patients Admitted to Intensive Care With COVID-19: Randomised Controlled Trial
Acronym: AZIQUINE-ICU
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Steering Committee decision in accordance with stopping rule 1: Emergence of new data
Sponsor: Frantisek Duska, MD, PhD (Other)
Collaborators: Masaryk Hospital Usti nad Labem (Other); University Hospital Pilsen (Other); The Faculty Hospital Na Bulovce (Other); St. Anne's University Hospital Brno, Czech Republic (Other); University Hospital, Motol (Other); General University Hospital, Prague (Other); University Hospital Olomouc (Other)
Responsible Party: Sponsor-Investigator, Frantisek Duska, MD, PhD, Dr, Charles University, Czech Republic
Organization: Charles University, Czech Republic (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AZIQUINE-ICU-25032020; 2020-001456-18 (EudraCT Number)
Record Dates: First submitted 2020-04-06; First posted 2020-04-09 (Actual); Last update posted 2020-11-06 (Actual); Status verified 2020-11

CONDITIONS: COVID-19; Respiratory Failure
Keywords: covid-19; Azithromycin; Hydroxychloroquine; Respiratory failure; Intensive Care
MeSH Terms: conditions — COVID-19; Respiratory Insufficiency | interventions — Azithromycin; Hydroxychloroquine

STUDY DESIGN:
Intervention Model Description: Prospective, multi-centre, randomised, pragmatic, double blind trial
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Visually unrecognisable IP or placebo will be prepared by dedicated unblinded study pharmacist and handed over to care provider immediately before administration
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- HC-A group (Experimental): * Day 1: Patients receive two doses 400 mg of Hydrochloroquine in 12 hours interval and 500 mg of Azithromycin once in 24 hours (with the first dose of hydrochloroquine)
  * Days 2-5: Patients receive two doses 200 mg of Hydrochloroquine in 12 hours interval 250 mg of Azithromycin once in 24 hours (with the first daily dose of hydrochloroquine)
  Interventions: Drug: Azithromycin; Drug: Hydroxychloroquine
- HC group (Active Comparator): * Day 1: Patients receive two doses 400 mg of Hydrochloroquine in 12 hours interval and placebo once in 24 hours (with the first dose of hydrochloroquine)
  * Days 2-5: Patients receive two doses 200 mg of Hydrochloroquine in 12 hours interval and placebo once in 24 hours (with the first dose of hydrochloroquine)
  Interventions: Drug: Hydroxychloroquine; Drug: Placebo
- C group (Placebo Comparator): • Day 1-5: Patients receive two doses of placebo in 12 hours interval and 1 extra dose of placebo once in 24 hours
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Azithromycin — orally or into nasogastric tube for 5 days
  Arms: HC-A group
Drug: Hydroxychloroquine — orally or into nasogastric tube for 5 days
  Arms: HC group; HC-A group
Drug: Placebo — orally or into nasogastric tube for 5 days
  Other Names: aqua pro injectione
  Arms: C group; HC group

SUMMARY:
Trial design: Prospective, multi-centre, randomised, pragmatic, double blind trial

Methods:

Participants: Adult (>18 years) within 24 hours of admission to intensive care unit with proven or suspected COVID-19 infection, whether or not mechanically ventilated. Exclusion criteria: symptoms of febrile disease for ≥1 week, treatment limitations in place or moribund patients, allergy or intolerance of any study treatment, incl. long QT syndromes, participation in another outcome-based interventional trial within last 30 days, patients taking Hydrochloroquine for other indication than COVID-19, pregnancy.

Interventions: Patients will be randomised in 1:1:1 ratio to receive Hydrochloroquine 800mg orally in two doses followed by 400mg daily in two doses and Azithromycin 500 mg orally in one dose followed by 250 mg in one dose for a total of 5 days (HC-A group) or Hydrochloroquine+ placebo (HC group) or placebo + placebo (C-group) in addition to best standard of care, which may evolve during the trial period but will not differ between groups.

Objective: To test the hypothesis that early administration of combination therapy slows disease progression and improves mechanical-ventilation free survival.

Outcomes:

Primary outcome: Composite percentage of patients alive and not on end-of-life pathway who are free of mechanical ventilation at day 14.

Secondary outcomes:

Composite percentage of patients alive and not on end-of-life pathway who are free of mechanical ventilation at day 14 in the subgroup of patients without the need of mechanical ventilation at baseline.

ICU-LOS D28 and D 90 mortality (in hospital)

Tertiary (exploratory) outcomes:

Viral load at D7 of study enrolment (No of viral RNA copies/ml of blood), proportion of patients alive and rtPCR negative from nasal swab at D14, Difference of FiO2 requirement and respiratory system compliance between day 0 and 7.

Randomization: In 1:1:1 ratio and stratified according to study centre and patients age (cut-off 70 years) Blinding (masking): Patients, treating clinicians, outcome assessors and data analyst will be blinded to study treatment allocation. Unblinded study pharmacist or research nurse will prepare investigational products.

DETAILED DESCRIPTION:
Introduction Background and objectives. In early 2020 novel Coronavirus disease (COVID-19) begun to spread from Asia to Europe and beyond forcing WHO to declare global pandemic. Infected patients shed the virus for a median of 20 days. Up to 10% of COVID-19 infected patients develop a severe form of disease requiring intensive care admission and some of them die. SARS-Cov2 is encapsulated positive strand RNA virus that uses ACE-2 of type 2 pneumocytes as binding sites. It has been hypothesised (Gattinoni 2020 ICM editorial) that initial hypoxemia caused by loss of primary injury to pulmonary vasculature leads to hyperventilation and patients self-inflicted lung injury predominantly in lung areas of increase stress and strain. In turn, later during the course of the disease, ARDS develops with a typical restrictive pattern of a stiff, wet and recruitable lung. At presents there is no evidence-based causative treatment of SARS-CoV-2 and there is a burning need of randomised-controlled trials to find effective therapeutic strategies intervention.

Explanation of rationale: Chloroquine has been used for malaria treatment and chemoprophylaxis, and hydroxychloroquine is used for treatment of rheumatoid arthritis, systemic lupus erythematosus and porphyrias. Both drugs have in-vitro activity against SARS-CoV, SARS-CoV-2, and other coronaviruses, with hydroxychloroquine having relatively higher potency against SARS-CoV-2 known to be susceptible in vitro to exposure to Hydrochloroquine. At the moment clinical trials are ongoing to test clinical efficacy in pre- and post-exposure prophylaxis in SARS-CoV-2. In one highly cited French non-randomised observational study by Gautret et. al., a significant reduction of virus carriage has been observed in patients co-incidentally treated by Azithromycin in addition to Hydrochloroquine as a part of initial empirical therapy of community-acquired pneumonia. Azithromycin is a macrolide antibiotic, which binds to the 50S subunit of the bacterial ribosome, thus inhibiting translation of mRNA. The positive-sense RNA viruses and indeed all genes defined as positive-sense can be directly accessed by host ribosomes to immediately form proteins and the effects of Azithromycin on this process are not known. No data are available at present on the clinical efficacy of Hydrochloroquine alone or in combination with Azithromycin and it is likely that any treatment affecting virus replication would only be effective if administered early, before overt ARDS develops.

In the light of this, the investigators designed a trial in which a hypothesis is tested, that early administation of hydrochlorochine alone or in combination with azithromycin can prevent respiratory deterioration in patients admitted to intensive care due to rapidly progressive COVID-19 infection.

Methods Trial design: Prospective, multi-centre, randomised, pragmatic, double blind trial Participants: Eligibility criteria for participants: Adult (>18 years) within 24 hours of admission to intensive care unit with proven or suspected COVID-19 infection. For the purpose of this study, intensive care unit is defined as a facility that allow continuous monitoring of vital functions and oxygen administration . It is expected that most patients will have rtPCR test known within 24 hours of admission to hospital. Nonetheless, if this is not the case (eg. due to overloaded lab facility, lack of supplies) it is possible to randomise a patient based on a strong clinical suspicion of SARS-Cov-2 infection. In case COVID-19 is not confirmed in retrospect, experimental therapy is withdrawn and the study subject is withdrawn from "per protocol" analysis of the primary and secondary outcomes, but remains in "intention-to-treat" cohort for the analysis of safety. Exclusion criteria: symptoms of febrile disease for ≥1 week, pregnancy, treatment limitations in place or moribund patients, allergy or intolerance of any study treatment, incl. long QT syndromes, myasthenia gravis, allergies or known deficiency of glucose-6-phosphate dehydrogenase, participation in another outcome-based interventional trial within last 30 days, patients taking Hydrochloroquine for other indication than COVID-19.

Settings and locations: Central study site is FNKV University Hospital Prague, updated list of participating centres is listed in the appendix.

Interventions: Standard of care. All patients will receive best supportive care that will be monitored, but not protocolised. It is recognised that in the standard of care may substantially differ among study centres and that is why randomisation is stratified. The standard of care also may change in time during the course of the study, for example, if a new evidence emerges and changes the state-of-the art treatment recommendations. Any such event will trigger emergency steering committee meeting, and decision will be taken about further action. REB and regulatory authorities will be notified immediately about the decision taken.

Study medication: All study medication is provided as a kind gift of Zentiva, ltd. Unblinded study pharmacist will prepare into 40 mls of sterile water study medication, according to patient's allocation into the treatment arm:

* Hydrochloroquine sulphate 200mg
* Azithromycin dihydrate 500mg
* Lactose 500mg (Placebo)

See enclosed Specifications of Product characteristics. The medication will be administered in covered Jeannete syringe into nasogastric tube (for patients unable to swallowed) or drunk from a black mug by patients who are able to. In both cases at least 50 ml of water will be used for flush. Treatment group allocation is as follows:

STUDY GROUP HC-A Azithromycin Hydrochloroquine HC Lactose Hydrochloroquine C Lactose Lactose

Each study patient will be given:

* Day 1: Patients receive two doses 400 mg of Hydrochloroquine or placebo in 12 hours interval and 500 mg of Azithromycin or placebo once in 24 hours (with the first dose of hydrochloroquine or placebo)
* Days 2-5: Patients receive two doses 200 mg of Hydrochloroquine or placebo in 12 hours interval 250 mg of Azithromycin or placebo once in 24 hours (with the first dose of hydrochloroquine or placebo)

Adjusting IP administration to patients' swallowing capability and GI function:

During the study, 3 groups of patients will be enrolled. Those conscious and able to swallow will be given study medication in black mug to swallow. Patients unable to swallow with a nasogastric tube in place will be given the IP via the NG tube reconstituted in sterile water and flushed as per local NG medication guideline. Administration of the IP is temporarily omitted in patients who are unable to swallow but without NG access or do not tolerate any enteral intake (such as patients in profound shock). As soon as the condition preventing IP administration is eliminated, resumption of study medication follows the guidance for day 1.

Outcomes:

Primary outcome: Composite percentage of patients alive and not on end-of-life pathway who are free of mechanical ventilation at day 14.

Secondary outcomes:

Composite percentage of patients alive and not on end-of-life pathway who are free of mechanical ventilation at day 14 in the subgroup of patients without the need of mechanical ventilation at baseline.

ICU-LOS D28 and D 90 mortality

Tertiary (exploratory) outcomes:

Viral load at D7 (No of viral RNA copies/ml of blood), proportion of patients alive and rtPCR negative from nasal swab at D14, Difference of FiO2 ratio and respiratory system compliance between day 0 and 7.

Changes to trial outcomes after the trial commenced, with reasons: None at presents Sample size calculation: Based on data from Wuhan and Washington, where 67% of patients were dead in 2 weeks and half of the survivors needed protracted mechanical ventilation, the assumed incidence of the primary outcome in the control group (ie. being alive and off the ventilator in 2 weeks) to be 25%. The study gives us 80% chance to detect the increase of the primary outcome to 50% in one or both interventional groups at p<0.017 with 74 patients in each arm. In order to compensate for drop-out and low of follow up the plan is to enrol 240 subjects into the study. An interim analysis is planned after the primary outcome is known for the 120th subject.

Randomisation: Will be performed in blocks of 3 and stratified for study centre and age (above or at/below 70 years). Electronic Case Record Form (eCRF) will perform randomisation using random sequence script in software R and generates medication code. Rationale: Patient's age is single most powerful predictor of outcome and stratifying randomisation and stratification decreases probability of treatment groups being of different age at baseline by chance. In analogy, study centers may vary in the use of non-protocolised treatments, which could bias the results.

Implementation:

Prior to initiation of each centre, the central research coordinator will train the local dedicated study personnel in the use of e-CRF and other study procedures. The medication will be delivered in sealed numbered boxes and stored in ICUs. Adhering to Good Clinical Practice rules and guidelines is of upmost importance despite all the challenges during current pandemic situation. Nonetheless, the eCRF has been designed to balance the safe conduct of the clinical trial and feasibility of timely data entry during staff shortages and overload. In order to do so, all data that is not essential for safety can be input in retrospect.

Collection data on cointerventions. Data on interventions that the investigators know/think influence survival will be monitored and described. This include concomitant antiviral antimicrobial diagnosis. Data will also be collected on how the respiratory specimen for rtPCR diagnostic was collected (smear, endotracheal aspirate, bronchoalveolar lavage).

Statistical methods: Proportion of patients alive and off mechanical ventilation (primary outcome) between intervention and control groups will be calculated using chi square test. P-value is adjusted for multiple comparisons to p=0.017. Survival and ICU/length of stay will be compared using Kaplan-Maier's curves and exploratory analyses my multi-level regression in R. The plan is to analyse the primary outcome separately in patients who require mechanical ventilation at baseline from those who don't and in patients above or below 70 years of age as a priori subgroup analyses.

As mentioned above, primary and secondary outcomes will only be calculated in patients with confirmed COVID-19 infection who received at least one dose of IP. Adverse events will be calculated in all randomised patients (intention-to-treat analysis).

Ethical Considerations Benefits and risks. This trial investigates two drugs that are being used off label to treat patients with severe COVID-19 with a balance of potential benefits and harms. Potential benefit include good biological rationale and observational data to believe that one or both drugs can prevent progression of a disease which led to death in 67% of patients in similar condition to those in this study. Possible harms include QT prolongation and resulting life-threatening arrhythmias or retinopathy, which may result in blindness. The investigators believe that clinical equipoise regarding risk/benefit to individual patient justifies well the conduct of this RCT.

Informed consent procedure. Patients with decision-making capacity will be asked to provide written prospective informed consent (See Appendix I) to this protocol. It is expected that a significant proportion of screened patients will lack the capacity to provide informed consent due to altered consciousness, respiratory distress or sedation to facilitate mechanical ventilation. In this situation, the deferred consent policy will be applied as per local law: independent physician will confirm in writing that the patient lacks capacity and fulfils criteria. Then, patient himself/herself are approached to provide consent as soon as they regain capacity. They are given options to continue in the study, to withdraw with permission to use the data collected up to the point or to withdraw from the study and request deleting all data collected. Patient next of kin plays no formal role as surrogate decision maker as per Czech legislature. Nonetheless, the family will be informed when practical about their relative's enrolment into the trial and the family will be offered an information leaflet explaining the nature of the study. All serious adverse event that are suspected from being related to study interventions will be reposted to Research Ethics Board and regulatory authorities as per local legislation.

Stopping rules. All SUSARs will be reported to both REB and to the steering committee, who may decide to stop the trial for safety concerns. Apart from safety, other reasons for stopping the trial are:

1. Emergence of new data ( e.g. publication of the results of a big RCT) that may lead continuation of the trial unethical. This may be due to safety concerns of placebo group (in case strong clinical benefit is proven by other trial) or any of the interventional groups (e.g. if harm is reported by other trials). This rule also applies for emergence of a new treatment.
2. After interim analysis: The steering committee will review primary outcomes and the summary of adverse events in all 3 groups (labelled as A, B, C) whilst still blinded to treatment allocation. The treatment can be stopped if the following criteria are fulfilled:

   1. There is a significant difference in the primary outcome at p<0.017 in between the groups.
   2. Futility: The futility criterion is not binding for the steering committee. Based on available data the study statistician calculates the probability of being able to prove the null hypothesis with achieving the target number of subjects and the probability of type II error made by stopping the trial prematurely.
   3. Safety: In case the number of adverse events in one or more treatment groups is find uneven or unacceptably high.

Replication of key aspects of trial methods and conduct. The trial is designed to be fully reproducible in larger international multi-centre trial.

Role of the sponsors This is investigator-initiated trial endorsed by Czech Society of Anaesthesia and Intensive Care. The most significant resource for the study is unpaid voluntary work of all the personnel conducting the study, who decided to do so in times of worldwide pandemic crisis. Part of the resources were gathered from voluntary donors in a crowdfunding campaign conducted by medical student association. Pharmaceutical company Zentiva, ltd. was approached by investigators and kindly agreed to provide study medication at no cost; however, it has had nor will have any role in study design; collection, management, analysis, and interpretation of data; writing of the report; or the decision to submit the report for publication.

Dissemination of Results: The investigators will submit the main results of the trial in an open-access peer-reviewed journal within 3 months after 240th subject completed the 90-day follow up visit, which is expected to happen in Q4 of 2021. The investigators will make fully de-identified record-level raw data available in a public database.

Trial status: NOT YET RECRUITING (as of 1st April 2020)

Declarations:

The trial design is in accordance with Declaration of Helsinky and the protocol, care report form and informed consent formularies were reviewed and approved by FNKV University Hospital Research Ethics Board ("Ethical Committee") on 1st April 2020 (decision number KH 14-00-2020).

ELIGIBILITY:
Inclusion Criteria:

* Adult (>18 years) within 24 hours of admission to intensive care unit with proven or suspected COVID-19 infection. For the purpose of this study, intensive care unit is defined as a facility that allow continuous monitoring of vital functions and oxygen administration . It is expected that most patients will have rtPCR test known within 24 hours of admission to hospital. Nonetheless, if this is not the case (eg. due to overloaded lab facility, lack of supplies) it is possible to randomise a patient based on a strong clinical suspicion of SARS-Cov-2 infection. In case COVID-19 is not confirmed in retrospect, experimental therapy is withdrawn and the study subject is withdrawn from "per protocol" analysis of the primary and secondary outcomes, but remains in "intention-to-treat" cohort for the analysis of safety.

Exclusion Criteria:

* symptoms of febrile disease for ≥1 week, pregnancy, treatment limitations in place or moribund patients, allergy or intolerance of any study treatment, incl. long QT syndromes, myasthenia gravis, allergies or known deficiency of glucose-6-phosphate dehydrogenase, participation in another outcome-based interventional trial within last 30 days, patients taking Hydrochloroquine for other indication than COVID-19.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2020-05-13 (Actual); Primary Completion 2020-11-04 (Actual); Study Completion 2020-11-04 (Actual)

PRIMARY OUTCOMES:
Proportion of alive patients free off mechanical ventilation | 14 days after enrolment
  Composite percentage of patients alive and not on end-of-life pathway who are free of mechanical ventilation at day 14.

SECONDARY OUTCOMES:
Proportion of patients who avoided the need of mechanical ventilation | 14 days
  Composite percentage of patients alive and not on end-of-life pathway who are free of mechanical ventilation at day 14 in the subgroup of patients without the need of mechanical ventilation at baseline.
ICU LOS | 28 days
  Length of stay in intensive care unit
Mortality28 | 28 days
  Proportion of patients who died by day 28
Mortality90 | 90 days
  Proportion of patients who died by day 90

CONTACTS AND LOCATIONS:
Locations (1):
- František Duška, Prague, Česká Republika, Czechia

IPD SHARING:
Plan to Share IPD: Yes
Deidentified record-level data will be shared in a public database
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: within 6 months of study completion
URL: http://mendeley.com

REFERENCES:
- [Background] Zhou F, Yu T, Du R, Fan G, Liu Y, Liu Z, Xiang J, Wang Y, Song B, Gu X, Guan L, Wei Y, Li H, Wu X, Xu J, Tu S, Zhang Y, Chen H, Cao B. Clinical course and risk factors for mortality of adult inpatients with COVID-19 in Wuhan, China: a retrospective cohort study. Lancet. 2020 Mar 28;395(10229):1054-1062. doi: 10.1016/S0140-6736(20)30566-3. Epub 2020 Mar 11. PMID 32171076
- [Background] Wang M, Cao R, Zhang L, Yang X, Liu J, Xu M, Shi Z, Hu Z, Zhong W, Xiao G. Remdesivir and chloroquine effectively inhibit the recently emerged novel coronavirus (2019-nCoV) in vitro. Cell Res. 2020 Mar;30(3):269-271. doi: 10.1038/s41422-020-0282-0. Epub 2020 Feb 4. No abstract available. PMID 32020029
- [Background] Colson P, Rolain JM, Lagier JC, Brouqui P, Raoult D. Chloroquine and hydroxychloroquine as available weapons to fight COVID-19. Int J Antimicrob Agents. 2020 Apr;55(4):105932. doi: 10.1016/j.ijantimicag.2020.105932. Epub 2020 Mar 4. No abstract available. PMID 32145363
- [Background] Yao X, Ye F, Zhang M, Cui C, Huang B, Niu P, Liu X, Zhao L, Dong E, Song C, Zhan S, Lu R, Li H, Tan W, Liu D. In Vitro Antiviral Activity and Projection of Optimized Dosing Design of Hydroxychloroquine for the Treatment of Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2). Clin Infect Dis. 2020 Jul 28;71(15):732-739. doi: 10.1093/cid/ciaa237. PMID 32150618
- [Background] Gautret P, Lagier JC, Parola P, Hoang VT, Meddeb L, Mailhe M, Doudier B, Courjon J, Giordanengo V, Vieira VE, Tissot Dupont H, Honore S, Colson P, Chabriere E, La Scola B, Rolain JM, Brouqui P, Raoult D. RETRACTED: Hydroxychloroquine and azithromycin as a treatment of COVID-19: results of an open-label non-randomized clinical trial. Int J Antimicrob Agents. 2020 Jul;56(1):105949. doi: 10.1016/j.ijantimicag.2020.105949. Epub 2020 Mar 20. PMID 32205204
- [Background] Wang D, Hu B, Hu C, Zhu F, Liu X, Zhang J, Wang B, Xiang H, Cheng Z, Xiong Y, Zhao Y, Li Y, Wang X, Peng Z. Clinical Characteristics of 138 Hospitalized Patients With 2019 Novel Coronavirus-Infected Pneumonia in Wuhan, China. JAMA. 2020 Mar 17;323(11):1061-1069. doi: 10.1001/jama.2020.1585. PMID 32031570
- [Background] Arentz M, Yim E, Klaff L, Lokhandwala S, Riedo FX, Chong M, Lee M. Characteristics and Outcomes of 21 Critically Ill Patients With COVID-19 in Washington State. JAMA. 2020 Apr 28;323(16):1612-1614. doi: 10.1001/jama.2020.4326. PMID 32191259
- [Derived] Duska F, Waldauf P, Halacova M, Zvonicek V, Bala J, Balik M, Benes J, Klementova O, Kozakova I, Kubricht V, Le Roy A, Vymazal T, Rehorova V, Cerny V; Czech Anaesthesia Clinical Trials and Audit Network. Azithromycin added to hydroxychloroquine for patients admitted to intensive care due to coronavirus disease 2019 (COVID-19)-protocol of randomised controlled trial AZIQUINE-ICU. Trials. 2020 Jul 8;21(1):631. doi: 10.1186/s13063-020-04566-x. PMID 32641163